CLINICAL TRIAL: NCT06408363
Title: Effectiveness of Sequential Eustachian Tube Maneuvers in Hyperbaric Oxygen Conditions: A Randomized Controlled Study
Brief Title: Effectiveness of Sequential Eustachian Tube Maneuvers in Hyperbaric Oxygen Conditions
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Hospital Felicio Rocho (Other)
Responsible Party: Principal Investigator, Alan Rodrigues de Almeida Paiva, Principal investigator, Hospital Felicio Rocho
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Prevention
Other Study IDs: 74381223500005125
Record Dates: First submitted 2024-04-18; First posted 2024-05-10 (Actual); Last update posted 2026-02-09 (Actual); Status verified 2025-06

CONDITIONS: Barotrauma;Ear; Tympanum; Perforation
Keywords: Barotrauma; Tympanic Membrane Perforation; Eustachian Tube; Hyperbaric Oxygenation
MeSH Terms: conditions — Tympanic Membrane Perforation; Barotrauma

STUDY DESIGN:
Who Masked: Investigator, Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Maneuver group (Experimental): Patients in the experimental group will receive detailed training and guidance on pressure equalization techniques and barotrauma prevention measures before undergoing treatment in a hyperbaric chamber. The specific maneuvers to be implemented are outlined below:
  Toynbee Maneuver: This maneuver involves swallowing with both the mouth and nose closed, thereby reducing the pressure in the nasopharynx and tympanic cavity.
  Unilateral Passive Valsalva Maneuver: This technique involves occluding one external nasal valve while performing a Valsalva maneuver on the opposite side.
  These maneuvers will be performed continuously during the compression phase of the hyperbaric chamber, every 30 minutes after reaching the desired pressurization level, and continuously during the decompression phase.
  Interventions: Behavioral: Maneuver group
- Standard treatment (No Intervention): Patients will receive the standard instructions for the hyperbaric chamber without specific guidance on performing equalization maneuvers.

INTERVENTIONS:
Behavioral: Maneuver group — These maneuvers for Eustachian tube opening will be performed continuously during the compression phase of the hyperbaric chamber, every 30 minutes after reaching the desired pressurization level, and continuously during the decompression phase.
  Arms: Maneuver group

SUMMARY:
Middle ear barotrauma represents the predominant complication associated with hyperbaric oxygen therapy, manifesting symptoms ranging from otalgia to tympanic membrane perforation. Several pressurization protocols have been proposed to reduce the incidence of this trauma, but barotrauma is still the main cause of poor adherence to hyperbaric therapy. Therefore, this study aims to evaluate the effectiveness of serial tubal opening maneuvers to prevent barotrauma in patients undergoing treatment in a hyperbaric chamber.

ELIGIBILITY:
Inclusion Criteria:

* Patient undergoing the first hyperbaric session.
* Understanding and properly carrying out equalization maneuvers

Exclusion Criteria:

* Patients who did not understand the equalization maneuvers
* Patients with specific contraindications to hyperbaric therapy
* Patients with acute middle ear or tympanic membrane disease

Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 100 (Estimated)
Dates: Start 2023-05-01 (Actual); Primary Completion 2026-12-01 (Estimated); Study Completion 2026-12-01 (Estimated)

PRIMARY OUTCOMES:
Incidence Reduction of Barotrauma | Until completion of the study, on average 10 months
  Patients performing Eustachian tube opening maneuvers will experience a lower incidence of barotrauma

CONTACTS AND LOCATIONS:
Locations (1):
- Hospital Felicio Rocho, Belo Horizonte, Minas Gerais, Brazil